CLINICAL TRIAL: NCT03100981
Title: Internet-delivered Mindfulness-Based Cognitive Therapy for Symptoms of Depression, Anxiety, and Stress Among Women Treated for Breast Cancer and Men Treated for Prostate Cancer - Effects and Mechanisms
Brief Title: Online Mindfulness for Women Treated for Breast Cancer and Men Treated for Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Karolinska Institutet (Other); Region Stockholm (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Krop & Sind; R87-A5432 (Other Grant/Funding Number: The Danish Cancer Society (preparation scholarship)); 7-12.0736 (Other Grant/Funding Number: The Danish Foundation TrygFonden); R113-A7015-14-S34 (Other Grant/Funding Number: The Danish Cancer Society (Knæk Cancer))
Record Dates: First submitted 2017-03-16; First posted 2017-04-04 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2018-10

CONDITIONS: Anxiety Depression; Breast Cancer Female; Prostate Cancer
Keywords: Mindfulness-Based Cognitive Therapy; Internet-delivered; Breast cancer; Prostate cancer; Survivors; Depression; Anxiety; Stress
MeSH Terms: conditions — Prostatic Neoplasms; Breast Neoplasms; Depression; Anxiety Disorders | interventions — Mindfulness-Based Cognitive Therapy; Therapeutics

STUDY DESIGN:
Intervention Model Description: After baseline assessment, participants will be randomly assigned to either the intervention or the control group. Both groups will receive online questionnaires at 5 weeks (midway), 10 weeks (post treatment) and 36 weeks (6 months follow-up) after baseline assessment.
  The intervention group receives a therapist phone call prior to enrollment in the internet-delivered treatment and then participates in 8 weeks of therapist-assisted internet-delivered Mindfulness-Based Cognitive Therapy. The internet-delivered treatment also comprises weekly distress measures, including suicide risk screening, and assessment of working alliance at week 2, 4, and 7 of the course.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Assessors performing introduction calls are masked in the sense that participants will not be randomized until after the introduction call. All questionnaires are completed as online surveys and are hence masked for group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-delivered MBCT (Experimental): The intervention group will immediately receive 8 weeks of therapist-assisted internet-delivered Mindfulness-Based Cognitive Therapy.
  Interventions: Behavioral: Internet-delivered Mindfulness-Based Cognitive Therapy
- Waitlist control (Other): The control group will be on a waiting list to participate in Internet-delivered MBCT after the 6-months follow-up time has passed.
  Interventions: Behavioral: Waitlist control

INTERVENTIONS:
Behavioral: Internet-delivered Mindfulness-Based Cognitive Therapy — Internet-delivered Mindfulness-Based Cognitive Therapy is a trainer-assisted course based on the manual for Mindfulness-Based Cognitive Therapy for depression. The course consists of 8 modules, one per week, for 8 weeks and one additional week for flexibility for the participants. In total 9 weeks with weekly written contact to the personal instructor.
  Each module has an overall theme with written theory, approximately 45 minutes of daily mindfulness practice and other daily assignments with the purpose of strengthening awareness in the everyday life.
  Other Names: Mindfulness-Based Cognitive Therapy; I-MBCT; MBCT
  Arms: Internet-delivered MBCT
Behavioral: Waitlist control — Participants in the control arm of the study will receive treatment as usual, which means that they are not offered interventions targeting psycho-social distress but also not prevented from participating in or seeking other psycho-social treatment during the course of the study.
  After the 6-months follow-up time has passed participants will get the opportunity to participate in 8 weeks of therapist-assisted internet-delivered Mindfulness-Based Cognitive Therapy, if the intervention is found efficient.
  Other Names: Treatment as usual
  Arms: Waitlist control

SUMMARY:
AIM: The aim of the present study is to investigate if Internet-delivered Mindfulness-Based Cognitive Therapy (I-MBCT) can reduce symptoms of depression and anxiety among women treated for breast cancer and men treated for prostate cancer compared to a treatment as usual control group. Furthermore, the effect of I-MBCT on symptoms of stress, insomnia, quality of life, and self-compassion and the potential mediating effect of working alliance and mindfulness will be explored. Finally, the cost-effectiveness of the I-MBCT intervention will be explored.

BACKGROUND: Symptoms of depression, anxiety, and stress are prevalent late-effects among cancer patients and -survivors. Mindfulness-based interventions aim at improving affect tolerance and emotion regulation, which could be of particular relevance for cancer patients and survivors, and MBCT has been shown efficacious in treating symptoms of depression, anxiety, and stress among cancer patients and survivors. However, the availability of face-to-face delivered MBCT is limited and hence using the internet to deliver MBCT may be a cost-effective way of increasing the accessibility of the intervention to vulnerable patients with limited resources.

METHODS: A total of 155 participants will be recruited from Department of Oncology and Department of Urology at Aarhus University Hospital and randomized to two groups: I-MBCT and a treatment-as-usual wait-list control group. Assessments will be conducted at pre-, midway and post intervention and at a 6- months follow-up.

DETAILED DESCRIPTION:
BACKGROUND

Symptoms of depression, anxiety, and stress is common among both cancer patients and cancer survivors and can lead to prolonged hospitalization, reduced quality of life, and deteriorate prognosis. In Mindfulness-Based Cognitive Therapy (MBCT) participants practice attention towards the present moment and acceptance of feelings and physical discomfort. This is in particular relevant for cancer patients and -survivors who often experience psychological symptoms connected to negative thoughts about the past and worries about the future.

MBCT is an 8-week group intervention and has shown to be effective in treating psychological distress in cancer survivors. Many cancer survivors experience challenges in following a group intervention because of health related reduced mobility and work- and family schedule conflicts, and hence it is relevant to investigate an internet-delivered alternative to MBCT.

I-MBCT is a manualized treatment for breast- and prostate cancer survivors, based on the manual for Mindfulness-Based Cognitive Therapy for depression. I-MBCT consist of 8 weeks of mindfulness practice combined with reading theory and supported by weekly text messages and answers from a therapist.

AIMS AND HYPOTHESES

In a randomized controlled trial the efficacy of 8-weeks I-MBCT for breast- and prostate cancer survivors will be investigated.

1. The primary aim of the study is to investigate if Internet-delivered Mindfulness-Based Cognitive Therapy (I-MBCT) will reduce symptoms of depression and anxiety among women treated for breast cancer and men treated for prostate cancer and that the effect is remained at 6 months after the treatment.
2. The secondary aim is to explore the effect of I-MBCT on symptoms of stress, insomnia, and quality of life.
3. Furthermore, the study aims to explore the potential mediating effect of working alliance, self-compassion, and mindfulness.
4. Finally, the cost-effectiveness of the I-MBCT intervention will be explored.

PARTICIPANTS AND PROCEDURES

A total of 155 breast- and prostate cancer survivors are consecutively recruited from Aarhus University Hospital, Denmark. Staff at the Outpatient Clinics at Department of Oncology and Department of Urology will screen patients for psychological distress at follow-up check-ups. If the patients indicates a moderate to high level of psychological distress, further information about the project will be given and patients can sign up for study enrollment.

Participants will after initial screening receive a phone call from a project staff to clarify if inclusion criteria are met. After informed consent all participants will fill out the online baseline questionnaire and then be randomized to either I-MBCT or a wait-list control group receiving treatment as usual in a ratio of 7:3 by means of a computer-generated randomization list.

Participants fill out online questionnaires at baseline, midway (after 5 weeks), post treatment (after 10 weeks) and at follow-up after 6 months.

The intervention group receive the 8-weeks of therapist-assisted I-MBCT which contains assessment of the Therapeutic Alliance at 2, 4, and 7 weeks after treatment onset.

The statistical evaluation of the effect I-MBCT compared to the waitlist control will be performed with Multilevel Linear Models and post-hoc tests. The possible mediating effects will be evaluated using Preacher & Hayes bootstrapping method. All analyses will be performed with a two-sided significance level of .05.

REGISTRATION DETAILS

The study record reported in ClinicalTrials.gov is completely consistent with the protocol approved by the Central Region Denmark Committee on Health Research Ethics before enrollment start. The study was registered in ClinicalTrials.gov after enrollment had started but before any data analysis was initiated.

ELIGIBILITY:
Inclusion Criteria:

* Man treated for prostate cancer or woman treated for breast cancer
* Active cancer treatment must have been completed (radiation therapy, operation and chemotherapy) within the past 5 years. Ongoing endocrine therapy is all right.
* A minimum score of 3 on anxiety and/or depression items from Symptom Check-List-8, subscale in Common Mental Disorder Questionnaire (SCL-8, CMDQ).
* Internet access on a daily basis
* Must have a cell phone

Exclusion Criteria:

* Cancer recurrence or ongoing cancer treatment.
* Problems with reading and/or understanding Danish
* Insufficient IT skills
* Severe mental illness causing problems with following the internet-delivered treatment, e.g. dementia, known psychotic disorder or developmental disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-02-24 (Actual); Primary Completion 2017-11-27 (Actual); Study Completion 2018-06-27 (Actual)

PRIMARY OUTCOMES:
Symptoms of Depression | Change from baseline until post treatment (10 weeks after baseline) and 6 months post treatment
  Change in symptoms of depression assessed by Beck Depression Inventory II (BDI-II)
Symptoms of Anxiety | Change from baseline until post treatment (10 weeks after baseline) and 6 months post treatment
  Change in symptoms of anxiety assessed by State-Trait Anxiety Inventory Form Y (STAI-S)

SECONDARY OUTCOMES:
Symptoms of Stress | Change from baseline until post treatment (10 weeks after baseline) and 6 months post treatment
  Change in symptoms of stress assessed by the Perceived Stress Scale (PSS)
Cost-Effectiveness | Change from baseline until post treatment (10 weeks after baseline) and 6 months post treatment
  Change in The Short Form Health Survey (SF-12+)

OTHER OUTCOMES:
Insomnia | Change from baseline until post treatment (10 weeks after baseline) and 6 months post treatment
  Change in symptoms of insomnia assessed by Insomnia Severity Index (ISI)
Self-compassion | Change from baseline until post treatment (10 weeks after baseline) and 6 months post treatment
  Change in Self-compassion assessed by The Self-Compassion Scale (SCS)
Quality of Life | Change from baseline until post treatment (10 weeks after baseline) and 6 months post treatment
  Change in Quality of Life assessed by the World Health Organization Well-being index (WHO-5)

CONTACTS AND LOCATIONS:
Overall Officials: Eva R Nissen, MSc, Study Chair — University of Aarhus
Locations (1):
- Department of Psychology, Aarhus University, Aarhus, Central Region Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andersson G. Using the Internet to provide cognitive behaviour therapy. Behav Res Ther. 2009 Mar;47(3):175-80. doi: 10.1016/j.brat.2009.01.010. Epub 2009 Feb 20. PMID 19230862
- [Background] Cuijpers P, van Straten A, Andersson G. Internet-administered cognitive behavior therapy for health problems: a systematic review. J Behav Med. 2008 Apr;31(2):169-77. doi: 10.1007/s10865-007-9144-1. PMID 18165893
- [Background] Cook JE, Doyle C. Working alliance in online therapy as compared to face-to-face therapy: preliminary results. Cyberpsychol Behav. 2002 Apr;5(2):95-105. doi: 10.1089/109493102753770480. PMID 12025884
- [Background] Christensen S, Zachariae R, Jensen AB, Vaeth M, Moller S, Ravnsbaek J, von der Maase H. Prevalence and risk of depressive symptoms 3-4 months post-surgery in a nationwide cohort study of Danish women treated for early stage breast-cancer. Breast Cancer Res Treat. 2009 Jan;113(2):339-55. doi: 10.1007/s10549-008-9920-9. Epub 2008 Feb 16. PMID 18278553
- [Background] O'Connor M, Christensen S, Jensen AB, Moller S, Zachariae R. How traumatic is breast cancer? Post-traumatic stress symptoms (PTSS) and risk factors for severe PTSS at 3 and 15 months after surgery in a nationwide cohort of Danish women treated for primary breast cancer. Br J Cancer. 2011 Feb 1;104(3):419-26. doi: 10.1038/sj.bjc.6606073. Epub 2011 Jan 11. PMID 21224851
- [Background] Stanton AL. Psychosocial concerns and interventions for cancer survivors. J Clin Oncol. 2006 Nov 10;24(32):5132-7. doi: 10.1200/JCO.2006.06.8775. PMID 17093275
- [Background] Dalton SO, Laursen TM, Ross L, Mortensen PB, Johansen C. Risk for hospitalization with depression after a cancer diagnosis: a nationwide, population-based study of cancer patients in Denmark from 1973 to 2003. J Clin Oncol. 2009 Mar 20;27(9):1440-5. doi: 10.1200/JCO.2008.20.5526. Epub 2009 Feb 17. PMID 19224839
- [Background] Reich M, Lesur A, Perdrizet-Chevallier C. Depression, quality of life and breast cancer: a review of the literature. Breast Cancer Res Treat. 2008 Jul;110(1):9-17. doi: 10.1007/s10549-007-9706-5. Epub 2007 Aug 3. PMID 17674188
- [Background] Osborn RL, Demoncada AC, Feuerstein M. Psychosocial interventions for depression, anxiety, and quality of life in cancer survivors: meta-analyses. Int J Psychiatry Med. 2006;36(1):13-34. doi: 10.2190/EUFN-RV1K-Y3TR-FK0L. PMID 16927576
- [Background] Holm LV, Hansen DG, Johansen C, Vedsted P, Larsen PV, Kragstrup J, Sondergaard J. Participation in cancer rehabilitation and unmet needs: a population-based cohort study. Support Care Cancer. 2012 Nov;20(11):2913-24. doi: 10.1007/s00520-012-1420-0. Epub 2012 Mar 14. PMID 22415608
- [Background] Hofmann SG, Sawyer AT, Witt AA, Oh D. The effect of mindfulness-based therapy on anxiety and depression: A meta-analytic review. J Consult Clin Psychol. 2010 Apr;78(2):169-83. doi: 10.1037/a0018555. PMID 20350028
- [Background] Piet J, Wurtzen H, Zachariae R. The effect of mindfulness-based therapy on symptoms of anxiety and depression in adult cancer patients and survivors: a systematic review and meta-analysis. J Consult Clin Psychol. 2012 Dec;80(6):1007-20. doi: 10.1037/a0028329. Epub 2012 May 7. PMID 22563637
- [Background] Wurtzen H, Dalton SO, Elsass P, Sumbundu AD, Steding-Jensen M, Karlsen RV, Andersen KK, Flyger HL, Pedersen AE, Johansen C. Mindfulness significantly reduces self-reported levels of anxiety and depression: results of a randomised controlled trial among 336 Danish women treated for stage I-III breast cancer. Eur J Cancer. 2013 Apr;49(6):1365-73. doi: 10.1016/j.ejca.2012.10.030. Epub 2012 Dec 19. PMID 23265707
- [Background] Khoury B, Lecomte T, Fortin G, Masse M, Therien P, Bouchard V, Chapleau MA, Paquin K, Hofmann SG. Mindfulness-based therapy: a comprehensive meta-analysis. Clin Psychol Rev. 2013 Aug;33(6):763-71. doi: 10.1016/j.cpr.2013.05.005. Epub 2013 Jun 7. PMID 23796855
- [Background] Ljotsson B, Falk L, Vesterlund AW, Hedman E, Lindfors P, Ruck C, Hursti T, Andreewitch S, Jansson L, Lindefors N, Andersson G. Internet-delivered exposure and mindfulness based therapy for irritable bowel syndrome--a randomized controlled trial. Behav Res Ther. 2010 Jun;48(6):531-9. doi: 10.1016/j.brat.2010.03.003. Epub 2010 Mar 16. PMID 20362976
- [Background] Andersson G, Paxling B, Wiwe M, Vernmark K, Felix CB, Lundborg L, Furmark T, Cuijpers P, Carlbring P. Therapeutic alliance in guided internet-delivered cognitive behavioural treatment of depression, generalized anxiety disorder and social anxiety disorder. Behav Res Ther. 2012 Sep;50(9):544-50. doi: 10.1016/j.brat.2012.05.003. Epub 2012 May 18. PMID 22728647
- [Background] Spek V, Cuijpers P, Nyklicek I, Riper H, Keyzer J, Pop V. Internet-based cognitive behaviour therapy for symptoms of depression and anxiety: a meta-analysis. Psychol Med. 2007 Mar;37(3):319-28. doi: 10.1017/S0033291706008944. Epub 2006 Nov 20. PMID 17112400
- [Background] Baer, R. A. (2003), Mindfulness Training as a Clinical Intervention: A Conceptual and Empirical Review. Clinical Psychology: Science and Practice, 10: 125-143. doi:10.1093/clipsy.bpg015
- [Background] Bartley, T. Mindfulness-Based Cognitive Therapy for Cancer. (Wiley-Blackwell, 2012)
- [Background] Segal, Z. V., Williams, J. M. G. & Teasdale, J. D. Mindfulness-Based Cognitive Therapy for Depression. (The Guilford Press, 2013).
- [Background] Beck, A. T., Steere, R. A. & Brown, G. . Manual for the revised Beck Depression Inventory. (The Psychological Corporation, 1996)
- [Background] Gorsuch, R. L., Lushere, R. E. & Alto, P. State-Trait Anxiety Inventory. Prof. Psychol. 3, 389-390 (1971)
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Neff, K. D. The Development and Validation of a Scale to Measure Self-Compassion. Self Identity 2, 223-250 (2003)
- [Background] Horvath, A. O. & Greenberg, L. S. Development and validation of the Working Alliance Inventory. J. Couns. Psychol. 36, 223-233 (1989)
- [Background] Baer RA, Smith GT, Lykins E, Button D, Krietemeyer J, Sauer S, Walsh E, Duggan D, Williams JM. Construct validity of the five facet mindfulness questionnaire in meditating and nonmeditating samples. Assessment. 2008 Sep;15(3):329-42. doi: 10.1177/1073191107313003. Epub 2008 Feb 29. PMID 18310597